## CONSENT FORM FOR PARTICIPANTS IN RESEARCH PROJECTS





| | le of project: A Trial Exploring User Engagement with a Syrepression (RADAR: Engage) | nptom-Tracking Syste | em for |
|---|---|---|---|
| Etl | nical review reference number: | Version number: v3.0 | 11/03/21 |
| | | | Please<br>initial<br>box |
| 1. | I confirm that I have read and understood the information sheet dated 11/03/2021 (Version 3.0) for the above project. I have had the opportunity to consider the information and asked questions which have been answered to my satisfaction. | | |
| 2. | I consent voluntarily to be a participant in this project and understand that I can refuse to take part and can withdraw from the project at any time, without having to give a reason, up until 09/08/2021 | | |
| 3. | I consent to the processing of my personal information for the purposes explained to me in the Information Sheet. I understand that such information will be handled in accordance with the terms of the General Data Protection Regulation (GDPR) and the UK Data Protection Act 2018. | | |
| 4. | I understand that my information may be subject to review by refrom King's College London for monitoring and audit purposes. | esponsible individuals | |
| 5. | I understand that confidentiality and anonymity will be maintained, and it will not be possible to identify me in any research outputs | | |
| 6. | I give permission for the researcher to access my data from the of Depression and Relapse (RADAR) study that I previously part to be linked to data in the current study. | | |
| 7. | I give permission for the researcher to write to my GP if circums | stances require it. | |
| 8. | I consent to any interviews conducted during the study period be to my data being shared with a third-party transcriber who will he confidentiality agreement. I understand that I can refuse to particular interview without it impacting my participation in the rest of the state. | ave signed a<br>icipate in any study | |
| 9. | I agree to my anonymised data and quotes contributing to public outputs. | | |
| 10 | I agree that the researcher may use my data for future research shared anonymously with other researchers. I understand that a identifiable data would be reviewed and approved by a research | any such use of | |

| Name of Participant | Date | Signature |
|---|---|---|
| | e in future studies of a s | |
| , , , , , | - | retain my contact details so that I may ondon researchers who would like to |
| the results of the rese | | to, and now to get information about |
| 1 11 I know how to contact | t the researcher if I need | to, and how to get information about |